CLINICAL TRIAL: NCT04273945
Title: A Phase 3, Prospective, Multicenter, Double-blind, Double-dummy, Randomized, Active-controlled, Parallel-group, Group-sequential, Adaptive, Event-driven Study to Compare Efficacy, Safety, and Tolerability of Macitentan 75 mg Versus Macitentan 10 mg in Patients With Pulmonary Arterial Hypertension, Followed by an Open-label Treatment Period With Macitentan 75 mg
Brief Title: Outcome Study Assessing a 75 Milligrams (mg) Dose of Macitentan in Patients With Pulmonary Arterial Hypertension
Acronym: UNISUS
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Actelion (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CR108740; AC-055-315 (Other: Janssen Research & Development, LLC); 2019-002533-11 (EudraCT Number); 2024-515669-32-00 (Registry Identifier: EUCT number)
Record Dates: First submitted 2020-01-31; First posted 2020-02-18 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Pulmonary Arterial Hypertension
MeSH Terms: conditions — Pulmonary Arterial Hypertension | interventions — macitentan

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Macitentan 10 milligrams (mg) + Placebo (Active Comparator): Run-in period:Participants who are either endothelin receptor antagonist (ERA)-naïve or who are receiving daily dose of macitentan or ambrisentan less (<) 10 milligrams (mg), or daily dose of bosentan <250 mg, will enter 4-week open-label run-in period with macitentan 10 mg prior to randomization. ERA-pre-treated participants will bypass run-in period and will be randomized to either macitentan 75 mg or macitentan 10 mg directly.Double-blind Treatment (DBT) Period:Participants will receive macitentan 10 mg orally up to End of DBT.To maintain blind, participants will receive macitentan 37.5 mg-matching placebo for 4 weeks and macitentan 75 mg-matching placebo thereafter up to DBT.Treatment Extension Period:After EDBT, participants will receive macitentan 37.5 mg once a day (qd) orally for 4 weeks, prior to receiving open-label macitentan 75 mg qd orally for 2 years. To maintain blind, participants will receive macitentan 75 mg-matching placebo during 4-week uptitration.
  Interventions: Drug: Macitentan 10 mg; Drug: Macitentan 37.5 mg; Drug: Macitentan 75 mg; Drug: Placebo
- Macitentan 75 mg + Placebo (Experimental): Run-in period:Participants who are either ERA-naive or who are receiving a daily dose of macitentan or ambrisentan <10 mg, or a daily dose of bosentan <250 mg, will enter 4-week open-label run-in period with macitentan 10 mg prior to randomization. ERA-pre-treated patients will bypass the run-in period and will be randomized to either macitentan 75 mg or macitentan 10 mg directly.DBT Period: participants will receive macitentan 37.5 mg orally for 4 weeks and macitentan 75 mg thereafter up to End of DBT. To maintain the blind, participants will receive macitentan 10 mg-matching placebo up to End of DBT.Treatment Extension Period: After EDBT, participants will continue to receive macitentan 75 mg orally for 2 years. To maintain the blind, participants will receive macitentan 37.5 mg-matching placebo during the 4-week up-titration period.
  Interventions: Drug: Macitentan 10 mg; Drug: Macitentan 37.5 mg; Drug: Macitentan 75 mg; Drug: Placebo

INTERVENTIONS:
Drug: Macitentan 10 mg — Participants will receive macitentan 10 mg film-coated tablets orally.
  Other Names: JNJ-67896062
Drug: Macitentan 37.5 mg — Participants will receive macitentan 37.5 mg film-coated tablets orally.
  Other Names: JNJ-67896062
Drug: Macitentan 75 mg — Participants will receive macitentan 75 mg film-coated tablets orally.
  Other Names: JNJ-67896062
Drug: Placebo — Participants will receive matching placebo film-coated tablets orally.

SUMMARY:
The purpose of this study is to demonstrate superiority of macitentan 75 milligrams (mg) in prolonging the time to the first clinical events committee (CEC)-adjudicated morbidity or mortality (M/M) event in participants with symptomatic pulmonary arterial hypertension (PAH) compared to macitentan 10 mg.

ELIGIBILITY:
Inclusion Criteria:

* Target population: greater than or equal to (>=) 18 (or the legal age of consent in the jurisdiction in which the study is taking place) years of age
* Target population: Symptomatic Pulmonary Arterial Hypertension (PAH) in World Health Organization Functional Class (WHO FC) II, III, or IV
* Target population: PAH subtype falling in one of the below classifications: Idiopathic; Heritable; Drug- or toxin-induced; Related to: Connective tissue disease, HIV infection, Portal hypertension, and Congenital heart disease with small/coincidental cardiac defect with systemic-to-pulmonary shunt (for example atrial septal defect, ventricular septal defect, patent ductus arteriosus, atrioventricular septal defect) which does not account for the elevated pulmonary vascular resistance (PVR) or persistent PAH documented by an Right heart catheterization (RHC) >= 1 year after simple systemic-to pulmonary shunt repair
* PAH diagnosis confirmed by hemodynamic evaluation at rest at any time prior to screening: Mean pulmonary artery pressure (mPAP) greater than (>) 20 millimeters of mercury (mm Hg), and; Pulmonary artery wedge pressure (PAWP) or left ventricular end diastolic pressure (LVEDP) less than or equal to (<=) 15 mm Hg, and PVR >= 3 Wood Units (that is, >= 240 dyn*sec/cm^5)
* Able to perform the 6-minute walking test (6MWT) with a minimum distance of 50 meters (m) and maximum distance of 440m at screening. Participants able to walk more than 440m at screening are eligible if they are in WHO FC III or IV and n-terminal prohormone of brain natriuretic peptide or n-terminal pro B-type natriuretic peptide (NT-proBNP) level is >=300 nanograms per liter (ng/L) at screening, based on central laboratory results

Exclusion Criteria:

* Known presence of three or more of the following risk factors for heart failure with preserved ejection fraction at screening, based on records that confirm documented medical history: Body mass index (BMI) > 30 kilograms per meter square (kg/m^2), Diabetes mellitus of any type, Essential hypertension (even if well controlled); Coronary artery disease, that is, any of the following: history of stable angina, or known more than 50 percent (%) stenosis in a coronary artery, or history of myocardial infarction, or history of or planned coronary artery bypass grafting and/or coronary artery stenting
* Presence of moderate or severe obstructive lung disease (forced expiratory volume in 1 second [FEV1] / forced vital capacity [FVC] < 70%; and FEV1 < 60% of predicted after bronchodilator administration) ) in participants with a known or suspected history of significant lung disease as documented by a spirometry test performed within 1 year prior to screening
* Known moderate to severe hepatic impairment, defined as Child-Pugh Class B or C, based on records that confirm documented medical history
* Serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) > 1.5*upper limit of normal (ULN) at screening
* Hemoglobin < 100 gram per liter (g/L) (< 10 gram per deciliter [g/dL]) at screening

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 935 (Actual)
Dates: Start 2020-06-30 (Actual); Primary Completion 2025-10-07 (Actual); Study Completion 2029-02-20 (Estimated)

PRIMARY OUTCOMES:
Double-blind Treatment Period: Time to First Clinical Events Committee (CEC)-adjudicated Morbidity or Mortality (M/M) Events | Up to 4 years
  Time to first CEC-adjudicated M/M event on-treatment (ie.,up to 7 days after last dose of DB study intervention) is defined as time from randomization to first of following events: All-cause death, including death caused by on-treatment adverse event that occur within 4 weeks of study DB treatment discontinuation;non-planned Pulmonary Arterial Hypertension(PAH)-related hospitalization(including for worsening of PAH, atrial septostomy, lung transplantation with or without heart transplantation, or initiation of parenteral prostacyclins);PAH-related disease progression, defined as worsening of World Health Organization(WHO) Functional Class(FC) from baseline or deterioration by at least 15% in exercise capacity, as measured by 6-minute walk distance(6MWD), from baseline and confirmed by second 6MWD test performed on different day within 2 week of initial test or appearance or worsening of signs or symptoms of right-sided heart failure that require initiation of intravenous diuretics.

SECONDARY OUTCOMES:
Double-blind Treatment Period: Change From Baseline to Week 24 in 6MWD | Baseline up to Week 24
  The 6MWT is a non-encouraged test performed to quantify exercise tolerance and capacity. This standardized test measures the distance an individual is able to walk over a total of six minutes on a hard, flat surface. The goal is for the individual to walk as far as possible in six minutes.
Double-blind Treatment Period: Number of Participants with CEC-adjudicated Death due to PAH and/or Hospitalizations for PAH (First and Recurrent) Events on-treatment | Up to 4 years
  Number of Participants with CEC-adjudicated death or hospitalization due to PAH will be reported.
Double-blind Treatment Period: Change From Baseline to Week 24 in PAH Symptoms Based on PAH-SYMPACT Questionnaire- Cardiopulmonary Symptom Domain Score | Baseline up to Week 24
  The Cardiopulmonary Symptoms domain consists of 6 items reported on a 5-point Likert scale (from 0 to 4). The value 0 means "no symptom" and value 4 corresponds to "very severe symptoms". The symptoms part of the PAH symptoms and impact questionnaire (PAH-SYMPACT) is completed daily for a 7-day period. The recall period of symptom items is the last 24 hours. An average Cardiopulmonary Symptoms domain score is determined based on the daily scores of the 6 items.
Double-blind Treatment Period: Change From Baseline to Week 24 in PAH Symptoms Based on PAH-SYMPACT Questionnaire- Cardiovascular Symptom Domain Score | Baseline up to Week 24
  The Cardiovascular Symptoms domain consists of 5 items reported on a 5-point Likert scale (from 0 to 4). The value 0 corresponds to "no symptoms" and value 4 corresponds to "very severe symptoms". The symptoms part of the PAH-SYMPACT is completed daily for a 7 day period. The recall period of symptom items is the last 24 hours. An average cardiovascular symptoms domain score is determined based on the daily scores of the 5 items.
Double-blind Treatment Period: Time to Death Occurring Between Randomization and End of Double-blind Treatment (EDBT) | Up to 4 years
  Time to death occurring between randomization and EDBT will be reported.
Treatment Extension Period: Time to Death Occurring Between Randomization and End of Study (EOS) | Up to 6 years
  Time to death occurring between randomization and EOS will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Actelion Clinical Trials, Study Director — Actelion
Locations (274):
- United States (43):
  - Mayo Clinic, Phoenix, Arizona
  - Arizona Pulmonary Specialists, Ltd, Scottsdale, Arizona
  - Scripps Memorial Hospital, La Jolla, California
  - USC Keck, Los Angeles, California
  - Jeffrey S. Sager, MD Medical Corporation, Santa Barbara, California
  - Lundquist Institute for Biomedical Innovation at Harbor-UCLA Medical Center, Torrance, California
  - National Jewish Health, Denver, Colorado
  - Cleveland Clinic, Weston, Florida
  - Piedmont Healthcare, Atlanta, Georgia
  - Northside Hospital, Atlanta, Georgia
  - Advocate Christ Medical Center, Oak Lawn, Illinois
  - Indiana University, Indianapolis, Indiana
  - St. Vincent Medical Group, Inc., Indianapolis, Indiana
  - University Of Iowa - Hospitals & Clinics, Iowa City, Iowa
  - Norton Pulmonary Specialists, Louisville, Kentucky
  - Louisiana State University, New Orleans, Louisiana
  - University of Michigan, Ann Arbor, Michigan
  - Troy Beaumont, Troy, Michigan
  - Washington University School Of Medicine, St Louis, Missouri
  - Saint Louis University Academic Pavillion, St Louis, Missouri
  - University of Nebraska Medical Center, Omaha, Nebraska
  - Reno Heart Institute, Reno, Nevada
  - Winthrop University Hospital, Mineola, New York
  - Mount Sinai, New York, New York
  - Columbia University, New York, New York
  - Stony Brook University Medical Center, Stony Brook, New York
  - Duke, Durham, North Carolina
  - Lindner Clinical Trial Center/Christ Hospital, Cincinnati, Ohio
  - Integris Baptist Office, Oklahoma City, Oklahoma
  - The Oregon Clinic, Portland, Oregon
  - Oregon Pulmonary Clinic, Portland, Oregon
  - Oregon Health And Science University, Portland, Oregon
  - University of Pennsylvania, Philadelphia, Pennsylvania
  - Allegheny General Hospital of Research, Pittsburgh, Pennsylvania
  - Lankenau Medical Center, Wynnewood, Pennsylvania
  - AnMed Health, Anderson, South Carolina
  - UT Southwestern Medical Center, Dallas, Texas
  - Baylor College of Medicine (BCM) - Baylor Heart Clinic, Houston, Texas
  - Baylor Scott White - Plano, Plano, Texas
  - San Antonio Methodist TX Transplant Physicians Group, San Antonio, Texas
  - The Robert Larner, M.D. College of Medicine at The University of Vermont, Burlington, Vermont
  - University of Wisconsin Hospital and Clinics, Madison, Wisconsin
  - Medical College Of Wisconsin, Milwaukee, Wisconsin
- Argentina (8):
  - Sanatorio de la Trinidad Mitre, Buenos Aires
  - Sanatorio Guemes, C.a.b.a.
  - Hospital Italiano de Buenos Aires, Caba
  - Sanatorio Ramon Cereijo, Caba
  - Centro Médico Dra. De Salvo, Caba
  - Instituto de Cardiologia de Corrientes, Corrientes
  - Instituto Medico de La Fundacion Estudios Clinicos, Rosario
  - Instituto Cardiovascular de Rosario, Rosario
- Australia (7):
  - Flinders Medical Centre, Bedford Park
  - Royal Prince Alfred Hospital, Camperdown
  - The Prince Charles Hospital, Chermside
  - St Vincent's hospital, Darlinghurst
  - Royal Hobart Hospital, Hobart
  - Fiona Stanley Hospital, Murdoch
  - Westmead Hospital, Westmead
- Austria (3):
  - LKH-Univ. Klinikum Graz, Graz
  - Ordensklinikum Linz GmbH Elisabethinen, Linz
  - Medical University Vienna, Vienna
- Belarus (2):
  - The Republican Scientific-Practical Center ''Cardiology'', Minsk
  - Minsk Regional Clinical Hospital, Minsk
- Belgium (2):
  - ULB Hôpital Erasme, Brussels
  - UZ Leuven, Leuven
- Brazil (13):
  - Universidade Federal De Minas Gerais - Hospital das Clínicas, Belo Horizonte
  - Instituto das Pequenas Missionárias de Maria Imaculada - Hospital Madre Teresa, Belo Horizonte
  - Empresa Brasileira de Servicos Hospitalares-EBSERH-Hospital Universitario de Brasilia, Brasília
  - Sociedade Hospitalar Angelina Caron - Hospital Angelina Caron, Campina Grande do Sul
  - Ceti - Centro de Estudos Em Terapias Inovadoras, Curitiba
  - Ynova Pesquisa Clinica, Florianópolis
  - Universidade Federal de Goias - Hospital das Clinicas da UFG, Goiânia
  - Hospital das Clinicas de Porto Alegre, Porto Alegre
  - Uniao Brasileira de Educacao e Assistencia Hospital Sao Lucas da PUCRS, Porto Alegre
  - Instituto de Medicina Integral Professor Fernando Figueira, Recife
  - Fundacao do ABC Centro Universitario FMABC, Santo André
  - Secretaria de Estado da Saude Instituto Dante Pazzanese de Cardiologia, São Paulo
  - Hospital Das Clinicas Da Faculdade De Medicina Da USP, São Paulo
- Bulgaria (2):
  - Multiprofile Hospital For Active Treatment National Cardiology Hospital, Ead, Sofia
  - University Multiprofile Hospital for Active Treatment- UMHAT Sveta Anna AD, Sofia
- Canada (4):
  - St. Joseph's Health Centre, Hamilton, Ontario
  - University of Ottawa Heart Institute, Ottawa, Ontario
  - University Health Network - Toronto General Hospital, Toronto, Ontario
  - Jewish General Hospital, Montreal, Quebec
- China (14):
  - Beijing Chaoyang Hospital, Beijing
  - Beijing Anzhen Hospital, Beijing
  - Peking Union Medical College Hospital, Beijing
  - The Second Xiangya Hospital of Central South Hospital, Changsha
  - West China Hospital Sichuan University, Chengdu
  - The First Affiliated Hospital of Chongqing Medical University, Chongqing
  - The First Affiliated Hospital of Guangzhou Medical University, Guangzhou
  - Shanghai Pulmonary Hospital, Shanghai
  - Renji Hospital, Shanghai
  - Zhongshan Hospital Fudan University, Shanghai
  - The General Hospital of Northern Theater Command, Shenyang
  - Shengjing Hospital Of China Medical University, Shenyang
  - Tianjin Medical University General Hospital, Tianjin
  - The First Affiliated Hospital of Xian Jiaotong University, Xi'an
- Colombia (5):
  - Fundacion Neumologica Colombiana, Bogotá
  - Fundacion Cardiovascular de Colombia, Bucaramanga - Piedecuesta - Valle de Menzuli
  - Clínica Imbanaco S.A.S., Cali
  - Centro Cardiovascular Colombiano Clínica Santa María, Medellín
  - Hospital Universidad del Norte, Soledad
- General University Hospital II.department of Internal Medicine-cardiology and angiology, Prague, Czechia
- Århus Universitetshospital, Skejby, Hjertemedicinsk Afdeling B, Aarhus, Denmark
- France (8):
  - CHU de Brest - Hopital de la Cavale Blanche, Brest
  - Hôpital Côte de Nacre, Caen
  - Hopital Bicetre Aphp Hopitaux Universitaires Paris Sud, Le Kremlin-Bicêtre
  - CHRU de Lille Hopital Claude Huriez, Lille
  - Aphm - Hopital Nord, Marseille
  - Centre Hospitalier Universitaire - de Nice - Hopital Pasteur, Nice
  - CHU Saint Etienne Hopital Nord, Saint-Priest-en-Jarez
  - Hopital Larrey CHU de Toulouse, Toulouse
- Germany (4):
  - Ruhr Universitat Bochum Diabeteszentrum, Bad Oeynhausen
  - Medizinische Hochschule Hannover, Hanover
  - Medizinische Klinik und Poliklinik V Klinikum Grosshadern der LMU, München
  - Universitaetsklinikum Regensburg, Regensburg
- Greece (4):
  - University Hospital of Alexandroupolis, Alexandroupoli
  - Alexandra General Hospital of Athens, Athens
  - University Hospital Of Larissa, Larissa
  - Ahepa University General Hospital of Thessaloniki, Thessaloniki
- Hungary (4):
  - Semmelweis Egyetem,Pulmonológiai Klinika, Budapest
  - Gottsegen Gyorgy Orszagos Kardiovaszkularis Intezet Felnott kardiologiai osztaly, Budapest
  - Pecsi Tudomanyegyetem Altalanos Orvostudomanyi Kar, Pécs
  - Szegedi Tudományegyetem, Általános Orvostudományi Kar, Családorvosi Intézet és rendelő, Szeged
- India (13):
  - NHL Medical College (SVP Hospital IMSR), Ahmedabad
  - Cims Hospital, Ahmedabad
  - Narayana Hrudayalaya Limited, Bangalore
  - SRM Medical College Hospital & Research Centre, Chengalpetu
  - Govindaswamy Kuppuswamy Naidu Memorial Hospital, Coimbatore
  - HealthWorld Hospitals, Durgapur
  - Renova Century Hospitals, Hyderabad
  - Care Hospitals, Hyderbad
  - Rabindranath Tagore International Institute of Cardiac Sciences, Kolkata
  - GB Pant Institute of Post Graduate Medical Education & Research, New Delhi
  - Sir Ganga Ram Hospital, New Delhi
  - Jawaharlal Institute of Postgraduate Medical Education and Research, Puducherry
  - B.D. Mehta Mahavir Heart Institute, Surat
- Israel (5):
  - Carmel Medical Center, Haifa
  - Shaare Zedek Medical Center, Jerusalem
  - Kaplan Medical Center, Rehovot
  - The Chaim Sheba Medical Center, Tel Litwinsky
  - Yitzhak Shamir Medical Center, Ẕerifin
- Italy (6):
  - ASST Grande Ospedale Metropolitano Niguarda, Milan
  - AOU Di Modena Policlinico Di Modena, Modena
  - Ospedale San Francesco, Nuoro
  - Fondazione IRCCS Policlinico San Matteo, Pavia
  - Fondazione Toscana Gabriele Monasterio CNR, Pisa
  - Policlinico Gemelli Universita Cattolica, Roma
- Japan (23):
  - The University of Tokyo Hospital, Bunkyō City
  - Kyushu University Hospital, Fukuoka
  - Kure Kyosai Hospital, Hiroshima
  - Kagoshima University Hospital, Kagoshima
  - St Marianna University Hospital, Kanagawa
  - Kanazawa University Hospital, Kanazawa
  - Kobe University Hospital, Kobe
  - Kurume University Hospital, Kurume
  - University Hospital Kyoto Prefectural University of Medicine, Kyoto
  - Kyoto University Hospital, Kyoto
  - Shinshu University Hospital, Matsumoto
  - Nagasaki University Hospital, Nagasaki
  - Nagoya University Hospital, Nagoya
  - Nagoya City University Hospital, Nagoya
  - Niigata University Medical And Dental Hospital, Niigata
  - Okayama University Hospital, Okayama
  - National Hospital Organization Okayama Medical Center, Okayama
  - Sapporo Medical University Hospital, Sapporo
  - Hokkaido University Hospital, Sapporo
  - National Cerebral and Cardiovascular Center, Suita-Shi
  - Juntendo University Hospital, Tokyo
  - Fujita Health University Hospital, Toyoake
  - University of Tsukuba Hospital, Tsukuba
- Malaysia (4):
  - Hospital Pulau Pinang, George Town
  - Hospital Serdang, Kajang
  - Sarawak Heart Center, Kota Samarahan
  - Institut Jantung Negara (National Heart Institute), Kuala Lumpur
- Mexico (6):
  - Consultorio Privado del Dr. Gabriel Arturo Ramos Lopez, Guadalajara
  - Instituto Nacional de Cardiologia Dr. Ignacio Chavez, Mexico City
  - Operadora de Hospitales Angeles SA de CV Hospital Angeles Lomas, México
  - Hospital Universitario Dr Jose Eleuterio Gonzalez, Monterrey
  - Unidad de Investigacion Clinica en Medicina S.C. (UDICEM), Monterrey
  - Centro de Investigacion Clinica Chapultepec, Morelia
- Netherlands (4):
  - VUMC Amsterdam, Amsterdam
  - St. Antonius Ziekenhuis Nieuwegein, Nieuwegein
  - Radboud Umcn, Nijmegen
  - Erasmus MC, Rotterdam
- Norway (2):
  - Akershus Universitetssykehus, Nordbyhagen
  - Oslo University Hospital, Oslo
- Poland (8):
  - Uniwersytecki Szpital Kliniczny w Bialymstoku, Bialystok
  - Szpital Uniwersytecki nr 2 im dr Jana Biziela w Bydgoszczy, Klinika Kardiologii, Bydgoszcz
  - Uniwersyteckie Centrum Kliniczne, Gdansk
  - SPSK nr 7 SUM w Katowicach Gornoslaskie Centrum Medyczne im Prof Leszka Gieca, Katowice
  - Krakowski Szpital Specjalityczny im Jana Pawla II Oddzial Kliniczny Chorob Serca i Naczyn, Krakow
  - Uniwersytecki Szpital Kliniczny nr 2 PUM w Szczecinie, Szczecin
  - Panstwowy Instytut Medyczny Ministerstwa Spraw Wewnetrznych i Administracji, Warsaw
  - Wojewodzki Szpital Specjalistyczny we Wroclawiu Osrodek Badawczo Rozwojowy, Wroclaw
- Portugal (3):
  - Uls Coimbra - Hosp. Univ. Coimbra, Coimbra
  - Uls Sao Jose - Hosp. Santa Marta, Lisbon
  - Uls Santa Maria - Hosp. Pulido Valente, Lisbon
- Russia (10):
  - Altay Regional Cardiological Dispensary, Barnaul
  - Chelyabinsk Regional Clinical Hospital, Chelyabinsk
  - State Autonomous HealthCare Institution 'Interregional Clinical Diagnostic Center', Kazan'
  - Scientific and Research Institution of Cardiovascular Diseases Complex Problems, Kemerovo
  - Moscow City Clinical Hospital No.51, Moscow
  - National Medical Research Center of Cardiology of MoH of Russian Federation, Moscow
  - National medical Research Center n.a. V.A.Almazov of MoH of Russian Federation, Saint Petersburg
  - Samara Regional Clinical Cardiological Dispensary, Samara
  - State Autonomous Healthcare Institution of Tyumen Region 'Scientific and Practical Medical Center', Tyumen
  - Volgograd Regional Clinical Cardiology Center, Volgograd
- Saudi Arabia (2):
  - King Faisal Specialist Hospital & Research Center, Riyadh
  - King Fahad Medical City, Riyadh
- Serbia (2):
  - University Clinical Center of Serbia, Belgrade
  - Institute for Pulmonary Disease of Vojvodina, Kamenitz
- Singapore (2):
  - National University Heart Centre, Singapore, Singapore
  - National Heart Centre (NHC) Singapore, Singapore
- Slovakia (2):
  - Narodny ustav srdcovych a cievnych chorob, Bratislava
  - The Eastern Slovakia Institute of Cardiovascular Diseases, Košice
- South Africa (2):
  - Milpark Hospital, Johannesburg
  - Dr Kalla, Lenasia
- South Korea (4):
  - Severance Hospital Yonsei University Health System, Seoul
  - Asan Medical Center, Seoul
  - Samsung Medical Center, Seoul
  - Seoul National University Hospital, Seoul
- Spain (7):
  - Hosp Univ Vall D Hebron, Barcelona
  - Hosp. Del Mar, Barcelona
  - Hosp. Univ. 12 de Octubre, Madrid
  - Hosp. Univ. La Paz, Madrid
  - Hosp. Univ. Pta. de Hierro Majadahonda, Madrid
  - Hosp. Costa Del Sol, Málaga
  - Hosp Clinico Univ de Salamanca, Salamanca
- Sweden (2):
  - Sahlgrenska Universitetsjukhuset, Gothenburg
  - Skanes universitetssjukhus, Lund
- Taiwan (4):
  - National Cheng Kung University Hospital, Tainan
  - National Taiwan University Hospital, Taipei
  - Mackay Memorial Hospital, Taipei
  - Taipei Veterans General Hospital, Taipei
- Thailand (6):
  - Phramongkutklao Hospital and Medical College, Bangkok
  - Ramathibodi Hospital Mahidol University, Bangkok
  - Siriraj Hospital Mahidol University, Bangkok
  - Maharaj Nakorn Chiang Mai hospital Faculty of Medicine, Chiang Mai
  - Srinagarind Hospital, Khon Kaen University, Khon Kaen
  - Songklanagarind hospital, Songkhla
- Turkey (Türkiye) (16):
  - Adana City Hospital, Adana
  - Cukurova University Medical Faculty, Adana
  - Ankara Etlik Speciality Hospital, Ankara
  - Hacettepe University Medical Faculty, Ankara
  - Gazi University Medical Faculty, Ankara
  - Ankara Bilkent Sehir Hastanesi, Ankara
  - Akdeniz University Medical Faculty, Antalya
  - Bursa Yuksek Ihtisas Training and Research Hospital, Bursa
  - Pamukkale University Medical Faculty, Denizli
  - Siyami Ersek Training and Research Hospital, Istanbul
  - Marmara University Medical Faculty, Istanbul
  - Ege University Medical Faculty, Izmir
  - Tepecik Training and Research Hospital, Izmir
  - Dokuz Eylul University Medical Faculty, Izmir
  - Kartal Kosuyolu Yuksek Ihtisas Egitim Ve Arastirma Hastanesi, Kartal Istanbul
  - Mersin University Medical Faculty, Mersin
- Ukraine (8):
  - CNE 'Cherkasy Regional Cardiological Center of Cherkasy Regional Council', Cherkassy
  - Communal Noncommercial Enterprise Cherkasy Regional Hospital of Cherkasy Regional Council, Cherkasy
  - MI 'Dnipropetrovsk Regional Clinical Center of Cardiology and Cardiac Surgery', Dnipro
  - CNE' City Clinical Hospital #8' of Kharkiv City Council, Kharkiv
  - SI National Scientific Center Institute of Cardiology of M.D. Strazhesko of NAMS of Ukraine, Kyiv
  - State Institute Of Phthisiology And Pulmonology N.A. F.G. Yanovskiy Of Ams Ukraine, Kyiv
  - Communal Noncommercial Enterprise of Lviv Regional Council 'Lviv Regional Clinical Hospital', Lviv
  - Municipal Non-commercial Enterprise Ternopil University Hospital of Ternopil Regional Council, Ternopil
- United Kingdom (3):
  - Royal Free Hospital, London
  - Freeman Hospital, Newcastle upon Tyne
  - Sheffield Teaching Hospitals NHS Foundation Trust Royal Hallamshire Hospital, Sheffield
- Vietnam (5):
  - Hanoi Medical University Hospital, Hanoi
  - Cho Ray Hospital, Ho Chi Minh City
  - Tam Anh Hospital, Ho Chi Minh City
  - Tam Duc Heart Hospital, Ho Chi Minh City
  - University Medical Center Ho Chi Minh city, Ho Chi Minh City

IPD SHARING:
Plan to Share IPD: Yes
The data sharing policy of the Janssen Pharmaceutical Companies of Johnson & Johnson is available at www.janssen.com/clinical-trials/transparency. As noted on this site, requests for access to the study data can be submitted through Yale Open Data Access (YODA) Project site at yoda.yale.edu.
URL: https://www.janssen.com/clinical-trials/transparency